CLINICAL TRIAL: NCT06341686
Title: Efficacy and Safety of Prophylactic Use of Letermovir Versus Preemptive Strategy in Kidney Transplant Recipients at Higher Risk of Cytomegalovirus Infection: a Prospective Randomized Study
Brief Title: Evaluation of the Prophylactic Use of Letermovir in Kidney Transplant Recipients at Risk of Cytomegalovirus Infection
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital do Rim e Hipertensão (Other)
Responsible Party: Principal Investigator, Helio Tedesco Silva Junior, Investigador Principal, Hospital do Rim e Hipertensão
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 75471023.2.0000.0082
Record Dates: First submitted 2024-03-07; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: CMV Infection
Keywords: Cytomegalovirus; Letermovir; Kidney transplant
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — letermovir; Ganciclovir

STUDY DESIGN:
Intervention Model Description: 1. Patients randomized to the prophylaxis group: Letermovir 480mg, 1x/day, from D14 to D98. Letermovir prophylaxis will start on day 14 after the kidney transplant.
  2. Patients randomized to the preemptive treatment group: Preemptive treatment (PET) will begin on day 21, evaluating CMV DNAnemia weekly until D98.CMV DNAnemia weekly until day 98 (21, 28, 35, 42, 49, 56, 63, 70, 77, 84, 91 and 98). The threshold for starting treatment with Ganciclovir is a CMV DNAemiaDNAemia > 5,000 IU in a single measurement (CMV infection) OR any CMV DNAemia with any signs or symptoms associated with CMV (CMV syndrome or disease).
  3. In both groups, CMV DNAemia will be monitored weekly until day 98 (21, 28, 35, 42, 49, 56, 63, 70, 77, 84, 91 and 98), and after any acute rejection treatment occurring between 3 months and 6 months after kidney transplantation.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Letermovir (Experimental): Patients randomized to the prophylaxis group: Letermovir 480mg, 1x/day, from D14 to D98. Letermovir prophylaxis will start on day 14 after kidney transplantation. In both groups, CMV DNAemia will be monitored weekly until day 98 (21, 28, 35, 42, 49, 56, 63, 70, 77, 84, 91 and 98), and after any acute rejection treatment occurring between 3 months and 6 months after kidney transplantation.
  Interventions: Drug: Letermovir 480 MG
- Preemptive therapy (Active Comparator): Patients randomized to the preemptive treatment group:
  Preemptive treatment (PET) will begin on day 21, assessing CMV DNAnemia weekly until day 98 (21, 28, 35, 42, 49, 56, 63, 70, 77, 84, 91 e 98). The threshold for starting treatment with Ganciclovir is a CMV DNAemia > 5,000 IU in a single measurement (CMV infection). measurement (CMV infection) OR any CMV DNAemia with any signs or symptoms associated with CMV (syndrome or disease).c. In both groups, CMV DNAemia will be monitored weekly until day 98 (21, 28, 35, 42, 49, 56, 63, 70, 77, 84, 91 and 98), and after any acute rejection treatment occurring between 3 months and 6 months after kidney transplantation.
  Interventions: Drug: Ganciclovir

INTERVENTIONS:
Drug: Letermovir 480 MG — Oral Letermovir for 84 days is effective in the prophylaxis of CMV infection in high-risk kidney transplant recipients. Oral Letermovir for 84 days, is associated with a lower incidence of CMV infection in high-risk high-risk kidney transplant recipients. In addition, the use of Letermovir is safe and associated with a low incidence of CMV syndrome or disease up to 6 months after after kidney transplantation. Finally, prophylaxis with Letermovir is associated with a lower incidence of discontinuation of immunosuppressive drugs, reducing the risk of of clinical and subclinical acute rejection
  Arms: Letermovir
Drug: Ganciclovir — The threshold for starting treatment with Ganciclovir is a CMV DNAemia > 5,000 IU in a single measurement (CMV infection) measurement (CMV infection) OR any CMV DNAemia with any signs or symptoms associated with CMV (syndrome or disease).
  Arms: Preemptive therapy

SUMMARY:
The two main cytomegalovirus (CMV) prevention strategies are prophylaxis and preemptive therapy. Prophylaxis effectively prevents CMV infection after solid organ transplantation (SOT), but is associated with high rates of neutropenia and late onset of post-prophylactic disease. In contrast, preemptive therapy has the advantage of leading to lower rates of CMV disease and robust humoral and T-cell responses. It is widely used in hematopoietic cell transplant recipients, but is rarely used after solid organ transplant recipients due to logistical considerations.

DETAILED DESCRIPTION:
Oral Letermovir for 84 days is effective in the prophylaxis of CMV infection in high-risk kidney transplant recipients. Oral Letermovir for 84 days, is associated with a lower incidence of CMV infection in high-risk high-risk kidney transplant recipients. In addition, the use of Letermovir is safe and associated with a low incidence of CMV syndrome or disease up to 6 months after after kidney transplantation. Finally, prophylaxis with Letermovir is associated with a lower incidence of discontinuation of immunosuppressive drugs, reducing the risk of of clinical and subclinical acute rejection

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant or re-transplant recipients, aged ≥18 years;
* Undergoing induction therapy with anti-thymocyte globulin;
* Receiving maintenance treatment with Tacrolimus, Mycophenolate and Prednisone;
* Positive CMV serology for donor and recipient.

Exclusion Criteria:

* CMV serology positive for donor and negative for recipient;
* Multiple organ recipients, or other organs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-05 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of CMV syndrome or disease | 6 months after transplantation
  Proportion (%) of CMV syndrome or disease

SECONDARY OUTCOMES:
Incidence of patients with plasma CMV DNAemia > 200 IU | 3 months
  Proportion (%) of patients with plasma CMV DNAemia > 200 IU
Incidence of patients with CMV infection/syndrome/disease | 84 Days
  Proportion (%) of patients with CMV infection/syndrome/disease

CONTACTS AND LOCATIONS:
Overall Officials: Helio Tedesco, Principal Investigator — Doctor of Renal Transplant Unit

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kotton CN, Kumar D, Caliendo AM, Huprikar S, Chou S, Danziger-Isakov L, Humar A; The Transplantation Society International CMV Consensus Group. The Third International Consensus Guidelines on the Management of Cytomegalovirus in Solid-organ Transplantation. Transplantation. 2018 Jun;102(6):900-931. doi: 10.1097/TP.0000000000002191. PMID 29596116
- [Background] Henrique Pinto C, Tedesco-Silva H Jr, Rosso Felipe C, Nicolau Ferreira A, Cristelli M, Almeida Viana L, Aguiar W, Medina-Pestana J. Targeted preemptive therapy according to perceived risk of CMV infection after kidney transplantation. Braz J Infect Dis. 2016 Nov-Dec;20(6):576-584. doi: 10.1016/j.bjid.2016.08.007. Epub 2016 Sep 25. PMID 27643978
- [Result] de Paula MI, Bae S, Shaffer AA, Garonzik-Wang J, Felipe CR, Cristelli MP, Waldram MM, Massie AB, Medina-Pestana J, Segev DL, Tedesco-Silva H. The Influence of Antithymocyte Globulin Dose on the Incidence of CMV Infection in High-risk Kidney Transplant Recipients Without Pharmacological Prophylaxis. Transplantation. 2020 Oct;104(10):2139-2147. doi: 10.1097/TP.0000000000003124. PMID 31978003
- [Result] Felipe C, Ferreira AN, de Paula M, Viana L, Cristelli M, Medina Pestana J, Tedesco-Silva H. Incidence and risk factors associated with cytomegalovirus infection after the treatment of acute rejection during the first year in kidney transplant recipients receiving preemptive therapy. Transpl Infect Dis. 2019 Dec;21(6):e13106. doi: 10.1111/tid.13106. Epub 2019 Oct 29. PMID 31081566
- [Result] Felipe CR, Ferreira AN, Bessa A, Abait T, Ruppel P, Paula MI, Hiramoto L, Viana L, Martins S, Cristelli M, Aguiar W, Mansur J, Basso G, Silva Junior HT, Pestana JM. The current burden of cytomegalovirus infection in kidney transplant recipients receiving no pharmacological prophylaxis. J Bras Nefrol. 2017 Oct-Dec;39(4):413-423. doi: 10.5935/0101-2800.20170074. English, Portuguese. PMID 29319768
- [Result] Haidar G, Boeckh M, Singh N. Cytomegalovirus Infection in Solid Organ and Hematopoietic Cell Transplantation: State of the Evidence. J Infect Dis. 2020 Mar 5;221(Suppl 1):S23-S31. doi: 10.1093/infdis/jiz454. PMID 32134486
- [Result] Ljungman P, Boeckh M, Hirsch HH, Josephson F, Lundgren J, Nichols G, Pikis A, Razonable RR, Miller V, Griffiths PD; Disease Definitions Working Group of the Cytomegalovirus Drug Development Forum. Definitions of Cytomegalovirus Infection and Disease in Transplant Patients for Use in Clinical Trials. Clin Infect Dis. 2017 Jan 1;64(1):87-91. doi: 10.1093/cid/ciw668. Epub 2016 Sep 28. PMID 27682069
- [Result] Chemaly RF, Chou S, Einsele H, Griffiths P, Avery R, Razonable RR, Mullane KM, Kotton C, Lundgren J, Komatsu TE, Lischka P, Josephson F, Douglas CM, Umeh O, Miller V, Ljungman P; Resistant Definitions Working Group of the Cytomegalovirus Drug Development Forum. Definitions of Resistant and Refractory Cytomegalovirus Infection and Disease in Transplant Recipients for Use in Clinical Trials. Clin Infect Dis. 2019 Apr 8;68(8):1420-1426. doi: 10.1093/cid/ciy696. PMID 30137245